CLINICAL TRIAL: NCT02640703
Title: Effect of Morning vs. Evening Vaccination on Hypoxia and Bradycardia of Preterm Infants: a Randomised Controled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Christian Poets, Prof. Dr. med. Christian F. Poets, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Impfstudie
Record Dates: First submitted 2015-12-12; First posted 2015-12-29 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Premature Birth; Intermittent Hypoxiema
MeSH Terms: conditions — Premature Birth | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- morning vaccination (Active Comparator): Vaccination with Infanrix + Prevenar 13 between 7 and 10 am
  Interventions: Biological: Infanrix + Prevenar 13
- evening vaccination (Active Comparator): Vaccination with Infanrix + Prevenar 13 between 7 and 10 pm
  Interventions: Biological: Infanrix + Prevenar 13

INTERVENTIONS:
Biological: Infanrix + Prevenar 13 — Different time of application

SUMMARY:
Hypoxia/bradycardia are common symptoms after vaccination of preterm infants. Adults show diurnal variations in vaccination response, due to circadian regulation of the immune system. The investigators plan to investigate whether preterm infants also show differences in hypoxia/bradycardia rate upon morning vs. evening vaccination.

Hypoxia/bradycardia is recorded by pulse oximetry starting 24 hours before until 48 hours after vaccination; parents also kept a sleep-diary. 24 hours after vaccination interleukin-6, interleukin-1β and C-reactive protein get determined. To control vaccination response, pertussis- and haemophilus-titers are determined before vaccination and at 4 months corrected age.

DETAILED DESCRIPTION:
Intervention: First hexavalent vaccination given to very preterm infants either in the evening or in the morning.

Primary outcome: rate of desaturations (SpO2 <80%) and bradycardias (Pulse rate <100/min) in first 24 h following vaccination in evening vs. morning vaccination group Secondary outcomes: cytokine levels (IL 6, IL 1ß, CRP) measured 24 h after vaccination, pertussis- and haemophilus-titers as measured before and after vaccination, i.e. at 4 months corrected age, in evening vs. morning vaccination group

ELIGIBILITY:
Inclusion Criteria:

* gestational Age: 26+0 to 30+6 Weeks of gestational age

Exclusion Criteria:

* bronchopulmonary dysplasia
* periventricular leukomalacia
* intraventricular hemorrhage >°2
* congenital malformations

Ages: 30 Days to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of hypoxia and bradycardia events | 72 hours

SECONDARY OUTCOMES:
Vaccination titer in blood sample after vaccination compared to vaccination titer in blood sample before vaccination | Before vaccination and at the age of 4 months (corrected age)

CONTACTS AND LOCATIONS:
Overall Officials: Christian F. Poets, Prof., Principal Investigator — Dept. of Neonatology, Tuebingen University Hospital
Locations (1):
- University Childrens Hospital, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No